CLINICAL TRIAL: NCT00873418
Title: Coping Skills Training in Heart Failure: Outcomes and Mechanisms
Brief Title: Coping Skills and Heart Failure: Outcomes and Mechanisms
Acronym: COPE-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Pro00009707; 1R01HL091920-01A1 (NIH)
Record Dates: First submitted 2009-03-30; First posted 2009-04-01 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Heart Failure
Keywords: Heart Failure; Intervention; Cognitive Behavior Therapy; Quality of Life
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Coping Skills Training (Experimental): 16 week telephone intervention using coping skills training to teach heart failure patients self-management skills and how to cope more effectively with psychological distress associated with heart failure.
  Interventions: Behavioral: Coping skills training
- Educational Control (Active Comparator): 16 weekly telephone calls for extended (standardized) care on heart failure education.
  Interventions: Behavioral: Coping skills training

INTERVENTIONS:
Behavioral: Coping skills training — 16 weekly telephone session using to teach heart failure patients self-management skills and how to cope more effectively with psychological distress associated with heart failure.
  Other Names: COPE-HF

SUMMARY:
This study will evaluate whether heart failure patients receiving a 16 week telephone delivered, intervention using cognitive behavior therapy to facilitate self-management of heart failure will have better clinical outcomes than heart failure patients receiving a 16 week heart failure education intervention via telephone.

DETAILED DESCRIPTION:
Over 5 million Americans suffer from heart failure (HF), with an associated annual health care cost in excess of $33 billion. With 500,000 new cases developing each year, HF is the only major cardiovascular disease that is increasing in prevalence. Despite intensive medical therapy, symptom instability and clinical deterioration are common and lead to frequent physician visits, hospitalization, and ultimately death. HF symptoms, including dyspnea and fatigue, are a major source of distress for patients with HF, and often impose severe limitations on their daily activities. Depression also is common in HF patients, and its presence is associated with increased risk of hospitalization and mortality, independent of disease severity. There is growing evidence that behavioral management is a critical component of living with HF that can reduce hospitalizations and help optimize health status. Although previous studies have demonstrated that case-management programs are effective, benefits appear to be short-lived once ongoing care is reduced. Prior research from our laboratory and others has shown that coping skills training (CST), designed both to teach patients self-management skills and to cope more effectively with psychological distress associated with their medical condition, is effective for such chronic diseases as diabetes, ischemic heart disease, and lung disease. However, CST has not yet been evaluated as an intervention to facilitate self-management of HF. We propose a randomized clinical trial comparing a 16-week CST intervention with Extended (Standardized) Care in a study sample of 200 HF outpatients, who are receiving medical treatment for HF according to current clinical practice guidelines. The CST intervention, delivered over the telephone, is designed reduce stress and depression and to improve aspects of health behavior that are related to HF outcomes, including symptom monitoring, medication adherence, dietary compliance, and physical activity. Before and following treatment, patients will be carefully assessed on important intermediate medical endpoints including HF disease biomarkers (B-type natriuretic peptide, ejection fraction, vascular endothelial function, autonomic regulation, and inflammatory activity), as well as on quality of life (QoL) indicated by both physical and psychosocial functioning. Effects of CST on clinical outcomes will be evaluated according to all-cause hospitalizations or mortality over a median follow-up period of 3 years. The data generated by the proposed study will provide important insights regarding the value of CST over and above usual medical care. If successful, we believe that the study findings should translate into initial recommendations for the incorporation of CST into self-management behavioral interventions as cost-effective approaches to enhance disease management, QoL and longevity in HF patients.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 21 years or older
* New York Heart Association (NYHA) Class I-IV HF of at least 3-months duration
* Left ventricular Ejection Fraction (EF) < 40% by left ventricular angiography, nuclear wall motion study, or echocardiography, within 6 months of study enrollment
* Undergoing treatment with a stable medication regimen.

Exclusion Criteria:

* Myocardial Infarction (MI), Percutaneous Transluminal Coronary Angioplasty(PTCA), Coronary Artery Bypass Graft (CABG) within 3 months of enrollment
* HF due to correctable cause or condition such as uncorrected primary valvular disease
* Alcohol or drug abuse within 12 months
* Illness such as malignancies that are associated with a life-expectancy of < 12 months
* Current pregnancy
* Inability to provide informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2009-03; Primary Completion 2015-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Quality of Life, Heart Failure Disease Biomarkers and Clinical Outcomes | yearly
  The primary outcomes were: i) post intervention effects on HF disease biomarkers and QoL (both with alpha=0.01), and; ii) a composite measure of time to death or first hospitalization (with alpha=0.03) over a median follow-up period of 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Sherwood, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blumenthal JA, Zhu Y, Koch GG, Smith PJ, Watkins LL, Hinderliter AL, Hoffman BM, Rogers JG, Chang PP, O'Connor C, Johnson KS, Sherwood A. The modifying effects of social support on psychological outcomes in patients with heart failure. Health Psychol. 2019 Jun;38(6):502-508. doi: 10.1037/hea0000716. Epub 2019 Apr 18. PMID 30998063
- [Derived] Sherwood A, Blumenthal JA, Koch GG, Hoffman BM, Watkins LL, Smith PJ, O'Connor CM, Adams KF Jr, Rogers JG, Sueta C, Chang PP, Johnson KS, Schwartz J, Hinderliter AL. Effects of Coping Skills Training on Quality of Life, Disease Biomarkers, and Clinical Outcomes in Patients With Heart Failure: A Randomized Clinical Trial. Circ Heart Fail. 2017 Jan;10(1):e003410. doi: 10.1161/CIRCHEARTFAILURE.116.003410. PMID 28062537
- [Derived] Sherwood A, O'Connor CM, Routledge FS, Hinderliter AL, Watkins LL, Babyak MA, Koch GG, Adams KF Jr, Dupree CS, Chang PP, Hoffman BM, Johnson J, Bowers M, Johnson KS, Blumenthal JA. Coping effectively with heart failure (COPE-HF): design and rationale of a telephone-based coping skills intervention. J Card Fail. 2011 Mar;17(3):201-7. doi: 10.1016/j.cardfail.2010.11.001. Epub 2011 Jan 21. PMID 21362527